CLINICAL TRIAL: NCT06839521
Title: Development, Validity and Reliability of Android Based 6 Minute Walking Test
Brief Title: 6-Minute Walk Test Assessment Via Mobile App
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Prof. Dr., Izmir Democracy University
Other Study IDs: Android-35
Record Dates: First submitted 2025-02-05; First posted 2025-02-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Functional Capacity
Keywords: 6-Minute Walk Test; Android; Validity; Reliability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WalkTest-T: Traditional 6-minute walk test will be applied.
  Interventions: Other: Walk Test-T; Other: Walk Test-A
- Walk Test-A: Mobile application of 6-minute test will be applied.
  Interventions: Other: Walk Test-T; Other: Walk Test-A

INTERVENTIONS:
Other: Walk Test-T — 6MWT will be conducted according to traditional protocols. During the test, parameters such as heart rate, oxygen saturation, and walking distance will be measured and compared with traditional methods.
Other: Walk Test-A — In order to develop Android-based 6DYT, the system will be designed with a multidisciplinary team consisting of software engineer and physiotherapist. In this programme, separate algorithms will be developed for indoor and outdoor environments so that individuals can be evaluated in a hospital environment, at home or in daily life. In indoor environments, the GPS signal is lost or there is not enough signal strength. For this reason, the programme will be developed so that the gyroscope of the phone can be used for distance measurement. GPS signals will be used outdoors. In this way, the physical activity level of the individual both in the hospital and in daily life will be measured.

SUMMARY:
This study aims to develop an Android-based 6-Minute Walk Test (6MWT) application to facilitate quick and efficient functional capacity assessment in clinical settings. The project will be carried out by a multidisciplinary team of software engineers and physiotherapists, with algorithms developed for both indoor and outdoor environments. As GPS signals may be lost indoors, the program will utilize the phone's gyroscope for distance measurement, while GPS signals will be used outdoors. The study will include healthy individuals aged 18-65, without any exercise restrictions. Participants' demographic data will be recorded, and the 6MWT will be conducted according to traditional protocols. During the test, parameters such as heart rate, oxygen saturation, and walking distance will be measured and compared with traditional methods. The Android application will provide auditory and vibration cues at the start and end of the test and will report health data in real-time. The data will be presented as mean ± standard deviation for continuous variables, and the test reliability will be assessed using the test-retest method. Results will be reported as age- and gender-adjusted z-scores for objective functional decline.

DETAILED DESCRIPTION:
The 6-minute walk test (6MWT) is a widely used test for the objective assessment of functional exercise capacity in the management of patients with moderate to severe lung disease.Unlike pulmonary function testing, 6DYT captures the often coexisting extrapulmonary manifestations of chronic respiratory disease, including cardiovascular disease, frailty, sarcopenia and cancer. Unlike the cardiopulmonary exercise stress test, this test does not require complex equipment or technical expertise. In this low-complexity, safe test, the patient is asked to walk as far as possible along a 30 m corridor for a 6-min period, with the primary outcome measure being the 6-min walking distance in metres.In a healthcare setting, measurement of exercise capacity is important to understand a person's current status and to assess rehabilitation progress. The 6-minute walk test (6MWT), which measures the distance walked in 6 minutes, is a widely used clinical tool for this purpose. A smartphone with integrated sensors provides a suitable platform for wearable biomechanical applications. With a wearable system for 6DYT and minimal additional setup, additional information can be obtained and clinically useful and immediate output can be provided to assess physical function and gait characteristics without the need to purchase specialised medical equipment.Wearable sensors allow a person to walk freely at a self-selected and natural pace that is more representative of everyday life than some laboratory conditions.Many studies have used accelerometers to detect gait and calculate gait parameters such as cadence, step timing and symmetry. Accelerometers can also be used to assess physical activity levels in relation to 6DYT results.In a systematic review published in 2015, 47 applications related to smoking cessation, 7 applications related to hernia, 42 applications related to diabetes, 103 applications related to asthma, 19 applications related to personal health records, 69 applications related to HIV, 29 applications related to colorectal diseases, 46 applications related to cancer, 104 applications related to pain management and 26 applications related to bariatric surgery were used.When the literature was reviewed, studies on the android-based application of 6DYT were conducted, but no application was found in Android application markets. Therefore, the aim of our study is to develop an Android-based 6 Minute Walk Test and to investigate its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Not having a disease that prevents walking
* To be able to use a smartphone

Exclusion Criteria:

* Exercise restriction for any reason
* Pregnancy or any known cardiovascular, pulmonary, neurological, metabolic or haematological disease
* Having any problem that prevents communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted with healthy individuals.
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test | Before and up to 2 weeks
  Before and after the test, participants' height, body weight, resting heart rate, oxygen saturation, blood pressure, Borg Dyspnea, and fatigue levels are assessed. The test follows American Thoracic Society (ATS) guidelines in a 30-meter covered corridor. At the start and end, participants receive audible and vibration cues. The app notifies the remaining time, and pulse oximeter data is displayed in real time. The practitioner can monitor walking distance, heart rate, and oxygen saturation. At the end of the test, results are reported to both the participant and practitioner. Additional data, including step count, cadence, and step symmetry, are also calculated.
SpO2 | Before and up to 2 weeks
  In the evaluation, SpO2 will be measured with a Bluetooth pulse oximeter that sends synchronised information flow to the application at the beginning, middle, and end of 6 minutes. In addition, the application will report the average of the SpO2 obtained from the entire test.
Modified Borg Scale | Before and up to 2 weeks
  It is a scale commonly used to assess exertional dyspnoea severity and rest dyspnoea severity. It consists of ten items describing the severity of dyspnoea according to degrees. The fact that the severity of dyspnoea is defined in the Modified Borg Scale (MBS) makes it easier for patients to apply. In this scale, symptom intensity is displayed progressively in a 0-10 score, representing the "absence of dyspnea" and "maximum dyspnea" respectively. Higher scores mean a worse outcome.
Walking distance | Before and up to 2 weeks
  Walking distance measurement will be performed according to 6DYT protocols. It will also be compared with the data from the smartphone.
International Physical Activity Questionnaire - Short Form (IPA-SF) | Before and up to 2 weeks
  It is one of the most commonly used questionnaires to assess physical activity. Information can be collected by telephone, interview or self-administration. The short form is generally preferred because the long form is repetitive. The short form consists of seven questions and provides information about the time spent by the individual in sitting, walking, moderate and vigorous activities. The question types can vary from 'Last seven days' to 'Any week'.
Heart Rate | Before and up to 2 weeks
  In the evaluation, heart rate will be measured with a Bluetooth pulse oximeter that sends synchronised information flow to the application at the beginning, middle, and end of 6 minutes. In addition, the application will report the average heart rate obtained from the entire test.

CONTACTS AND LOCATIONS:
Overall Officials: Ferruh Taspinar, Prof. Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Betül TAŞPINAR, Konak, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No